CLINICAL TRIAL: NCT04232735
Title: Stimulating Evidence Based, Personalized and Tailored Information Provision to Improve Decision Making After Oesophagogastric CancEr Diagnosis - a Pragmatic Stepped Wedge Trial-
Brief Title: Evidence Based Information Provision to Improve Decision Making After Oesophagogastric Cancer Diagnosis (SOURCE)
Acronym: SOURCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W19_094#19.124
Record Dates: First submitted 2019-12-20; First posted 2020-01-18 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Oesophageal Cancer; Gastric Cancer
Keywords: Prediction models; Tailored information; Stepped Wedge Trial; Oesophageal cancer; Gastric cancer; Webtool; Health care provider training
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Pragmatic Stepped Wedge Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The Source tool is used by care givers for informing patients about the outcomes of treatment. Prediction models are developed and built in the website in order to generate a personalized prediction of the outcomes: survival, toxicity and/or complications and HRQL. These predictions are visualized in clear and comprehensible graphs with a broad variation of options available for tailoring of the visualizations.
  In order for care givers to be able to use this tool effectively, we designed the Source training. This communication skills training is comprised of an e-learning, two face-to-face group sessions and an individual booster session. Aside from an instruction video on the navigation within the Source tool, the e-learning consists of theory and tips and tricks on how to inform patients and communicate risks. The face-to-face components of the training are focused on getting the skilled use of the source tool into practice, by receiving personal feedback on the performance.
  Interventions: Other: Tool and training

INTERVENTIONS:
Other: Tool and training — The Source tool aims to assist health care providers with giving evidence based information about treatment outcomes by providing visualizations of personalized predictions of treatment outcomes for different treatments of oesophageal and gastric cancer. These predictions result from recently designed and updated prediction models on the survival, toxicity, complications and health related quality of life of oesophageal and gastric cancer patients.
  The training aims to teach participants to inform patients about outcomes of treatment. The training is placed in the context of shared decision making (SDM), following the 4-step model by Stiggelbout et al., 2015.8 The training is provided in small groups (3-6 participants) by an experienced trainer and supported by professional actors. The training aims to address knowledge, attitude and skills.

SUMMARY:
The overarching aim of the programme 'Stimulating evidence based, personalized and tailored information provision to improve decision making after oesophagogastric cancer diagnosis' (SOURCE) is to provide oesophagogastric cancer patients at all disease stages with evidence based and personalized information about survival, treatment-related side-effects and/or complications and health related quality of life, tailored to patients' specific information needs, to facilitate informed decision making about treatment and thereby optimize personal care and outcomes.

For this purpose the Source tool and training were designed. The Source tool is a prediction model based website to be used by care givers for informing patients about the outcomes of treatment. The Source training for care givers is designed to learn care givers how to inform patients effectively, especially about the outcomes of treatment.

DETAILED DESCRIPTION:
The overarching aim of the programme 'Stimulating evidence based, personalized and tailored information provision to improve decision making after oesophagogastric cancer diagnosis' (SOURCE) is to provide oesophagogastric cancer patients at all disease stages with evidence based and personalized information about survival, treatment-related side-effects and/or complications and health related quality of life, tailored to patients' specific information needs, to facilitate informed decision making about treatment and thereby optimize personal care and outcomes.

For this purpose the Source tool and training were designed. The Source tool is a prediction model based website to be used by care givers for informing patients about the outcomes of treatment. The Source training for care givers is designed to learn care givers how to inform patients effectively, especially about the outcomes of treatment.

The primary aim of the SOURCE trial is to investigate the effect of the tool and training on the (numerical) precision of information about outcomes of treatment in the treatment information consultation. Secondary outcomes include: patients' satisfaction, evaluation and knowledge of the information provided by the health care provider, evaluation of the decision made and health related quality of life.

A pragmatic stepped wedge design will be used to test the effect of intervention. 21 health care providers will include 3 patients as control measurements (before intervention) and 3 patients as intervention measurements (after intervention). Participating centers will be divided into geographical subgroups, in which the transition period (in which the intervention will take place) will be spread across time.

All oesophageal and gastric cancer patients scheduled for a treatment information consultation with a participating health care provider are suitable for inclusion and will be approached for participation in the SOURCE study. Measurements include audio recordings of the treatment information consultation and questionnaires filled in by patients and health care providers at different moments in time. Audio recordings will be scored and analyzed based on a study specific coding scheme.

The investigators estimate the physical burden/risk of this study to be negligible.

ELIGIBILITY:
Inclusion Criteria:

Health care providers:

* Specialist, physician assistant or nurse practitioner in the field of oncology, oncological radiotherapy or oncological surgery who are used to discussing treatment and treatment outcome with patients
* Informed consent for data collection
* Three audiorecorded treatment information consultations with oesophageal or gastric cancer patients before the scheduled transition period (control measurements)
* Three audiorecorded treatment information consultations with oesophageal or gastric cancer patients after the scheduled transition period (intervention measurements) and before the scheduled end date of the study

Patients:

* Age ≥ 18 years
* Histological or cytological proof of oesophageal or gastric cancer
* Informed consent for trial data collection A treatment information consultation with a participating doctor to discuss either curative treatment, first line palliative treatment, and/or best supportive care.

Exclusion Criteria:

Health care providers:

- Less than two control and/or intervention measurements

Patients:

* Cognitive impairment or insufficient understanding of the Dutch language
* GIST and smallcell carcinomas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
SOURCE observational scale | through study completion, an average of 1 year
  The SOURCE observational scale is developed to primary answer the following question: Does the combination of the tool and the training improve observed (numerical) precision of information about treatment outcomes in clinical consultations? Min. value: 1 Max. value:4 Higher scores mean higher (numerical) precision

SECONDARY OUTCOMES:
Continuing professional development (CPD) reaction Questionnaire | through study completion, an average of 1 year
  Health care providers' intention to inform patients about treatment outcomes using numbers (effect training only)
Patient Satisfaction Questionnaire (PSQ-5 patient and doctor version) | 2 weeks
  Patient and physician satisfaction with communication and decision making
Shared Decision Making Questionnaire (SDMQ-9) | 2 weeks
  Patient-reported shared decision making
Decisional Conflict Scale (DCS) | 2 weeks
  Patients' evaluation of the decision made
EORTC QLQ - INFO25 + tailor made items on treatment outcome information | 2 weeks
  Patients' evaluation and knowledge of the information provided by the health care provider
EORTC QLQ-C30 | 3 months vs. baseline
  Patients' health related quality of life, cancer specific
EORTC QLQ-OG25 | 3 months vs. baseline
  Patients' health related quality of life, gastro-intestinal cancer specific
Trust in the Oncologist Scale (TiOS-sf) | 2 weeks
  Patients' trust in the health care provider
State-Trait Anxiety Inventory (STAI) | 2 weeks vs. baseline
  Patients' anxiety
((Mini-)Mental Adjustment to Cancer scale ((Mini-)MAC) | 2 weeks vs. baseline
  Patients' helplessness/hopelessness + fighting spirit
Duration of consultation in minutes (min.) | through study completion, an average of 1 year
  Consultation time
Health care providers' personalization of treatment outcome information measured with SOURCE observational scale | through study completion, an average of 1 year
  Frequency of explicitly personalizing treatment outcome information, based on audio tapes Min. value: 0 Max. value: endless Higher values mean more utterances of personalization
Health care providers' tailoring of treatment outcome information measured with SOURCE observational scale | through study completion, an average of 1 year
  Frequency of explicitly tailoring treatment outcome information, based on audio tapes Min. value: 0 Max. value: endless Higher values mean more utterances of tailoring
Health care providers' use of visualizations of treatment outcome information measured with SOURCE observational scale | through study completion, an average of 1 year
  Frequency of explicitly showing visualizations treatment outcome information, based on audio tapes Min. value: 0 Max. value: endless Higher values mean more utterances of showing visualizations
Health care providers' use of time frames when giving treatment outcome information measured with SOURCE observational scale | through study completion, an average of 1 year
  Presence of time frame when giving treatment outcome information, in utterances coded for the primary outcome Min. value: 0 Max. value: 1 Value 1 means time frame present, value 0 means time frame absent
Treatment outcome category of health care providers' treatment outcome information measured with SOURCE observational scale | through study completion, an average of 1 year
  Treatment outcome category of health care providers' treatment outcome information, in utterances coded for the primary outcome Values: Survival, Health-related Quality of Life, Side effects and complications, Progression of tumor Non-ordinal variable
Person initializing treatment outcome information measured with SOURCE observational scale | through study completion, an average of 1 year
  Person taking the initaitive for the health care provider's treatment outcome information, in utterances coded for the primary outcome Values: Health care provider, Patient Non-ordinal variable
Health care providers' (numerical) precision of treatment outcome information measured with SOURCE observational scale simulated patient consultations (effect intervention) | through study completion, an average of 1 year
  Health care providers' (numerical) precision of treatment outcome information measured in simulated patient consultations (effect intervention) Min. value: 1 Max. value:4 Higher scores mean higher (numerical) precision

OTHER OUTCOMES:
Observed presence of Source tool measured with SOURCE observational scale | through study completion, an average of 1 year
  Health care providers' observed use of the Source tool Min. value: 0 Max. value:1 Value 0 means absence of Source tool in consultation, Value 1 means presence of Source tool in conversation
SOURCE evaluation questionnaire (tailor made evaluation questionnaire) | through study completion, an average of 1 year
  Health care providers' evaluation of the Source tool, training and e-learning Min value: 1 Max value: 10 Higher scores mean better evaluations

CONTACTS AND LOCATIONS:
Overall Officials: H WM van Laarhoven, Prof. Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (12):
- Netherlands (12):
  - Academic Medical Center, Amsterdam, North Holland
  - Flevoziekenhuis, Almere Stad
  - VUmc, Amsterdam
  - Radiotherapiegroep, Arnhem
  - Rijnstate, Arnhem
  - Catherina Ziekenhuis, Eindhoven
  - LUMC, Leiden
  - Maastro, Maastricht
  - Radboud UMC, Nijmegen
  - BVI, Tilburg
  - ETZ, Tilburg
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT04232735/Prot_000.pdf